CLINICAL TRIAL: NCT01215760
Title: Proposal of Sensory Reeducation in Peripheral Nerve Injuries of Median and Ulnar Nerves of the Hand: RANDOMIZED CONTROLLED CLINICAL STUDY
Brief Title: Sensory Reeducation in Peripheral Nerve Injuries of Hand
Acronym: HandtherRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Marisa de Cassia Registro Fonseca, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MFonseca
Record Dates: First submitted 2010-07-01; First posted 2010-10-06 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Median Nerve Disease; Ulnar Nerve Disease; Peripheral Nerve Disease
Keywords: peripheral nerve injury; sensory reeducation; brain plasticity; training with a mirror; rehabilitation
MeSH Terms: conditions — Median Neuropathy; Ulnar Neuropathies; Peripheral Nervous System Diseases; Peripheral Nerve Injuries | interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MIRROR (Active Comparator): Early sensory reeducation group, started at the first week postoperatively, using specific guidelines using the mirror training and stimulation of the contralateral side. Initially, the stimulation will be unilateral and later bilateral, after the removal of the splint in 4 weeks.
  Interventions: Other: Training with a mirror
- Home program (Active Comparator): The classical group iniciates after 16 weeks postoperatively and follow a standard home protocol for sensory reeducation. It begins with recognition of textures and objects, and specific rehabilitation, if any associated injuries.
  Interventions: Other: No mirror therapy

INTERVENTIONS:
Other: Training with a mirror — Early sensory reeducation group, started at the first week postoperatively, using specific guidelines using the mirror training and stimulation of the contralateral side. Initially, the stimulation will be unilateral and later bilateral, after the removal of the splint in 4 weeks.
  Other Names: Alternative stimuli for sensory reeducation; Mirror therapy; Home program
  Arms: MIRROR
Other: No mirror therapy — The classical group iniciates after 16 weeks postoperatively and follow a standard home protocol for sensory reeducation without the mirror. It begins with recognition of textures and objects, and specific rehabilitation, if any associated injuries.
  Other Names: home program; classic program; standard program
  Arms: Home program

SUMMARY:
Objectives: To develop a protocol for early treatment using sensory reeducation through the mirror after surgical reconstruction of the median nerve and / or ulnar hand, and its comparison with the evolution of the return of skin sensitivity after a not early rehabilitation which will be conducted by physiotherapists, with blinding of the evaluators.

DETAILED DESCRIPTION:
Changes in the cerebral cortex begins soon after peripheral nerve injury resulting in overlapping cortical areas on adjacent as a result of the absence of stimuli in the area of cortical representation of the injured nerve. Sensibility reeducation is a process of reprogramming the brain through a progressive learning proposing feed the somatosensory cortex with alternative stimulus to preserve the cortical map of the hand and facilitate the sensory recovery. This study is based on the hypothesis that sensory reeducation starting in the first days after surgery by training with the mirror promotes greater preservation of the cortical map of the original hand, with better functional results. We also believe that sensory reeducation performed early with the mirror will enhance the return of sensibility, emphasizing functional reorganization with less alteration of the cortical map of the hand. Metodology: Will be included patients over 18 with injury of the median and/or ulnar nerve at the first week after surgery. Patients will be randomized into an early group with the use of mirror and a classic group of sensory reeducation. In evaluating the Rosen score will be used with motor, sensory and pain/discomfort components. The assessment instruments used were: Semmes Weinstein monofilaments, Jamar® and Pinch Gauge® dynamometer, goniometry, shape and texture identification (STI), Sollerman test, Disabilities of the arm, shoulder and hand questionnaire (DASH), two points discriminator and numeric pain scale.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years
* male or female
* reconstruction of peripheral nerve or ulnar median
* primary or secondary graft through the Hospital of the Medical School of Ribeirão Preto, University São Paulo
* possible associated tendon and skin lesions
* flexor zones I, II, III, IV or V.

Exclusion Criteria:

* nerve damage that may associated with multiple complex lesions, bone or joint injuries
* presence of central nervous system injury
* chronic diseases metabolic and degenerative rheumatic diseases, leprosy and diseases affecting the peripheral nervous system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-03; Primary Completion 2010-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
sensory threshold | 1 month
  Semmes Weinstein monofilaments

SECONDARY OUTCOMES:
sensory threshold, range of motion, pain, function, tactile gnosia, pinch and grip strength | 3 months
  Semmes Weinstein monofilaments, Jamar® and Pinch Gauge® dynamometer, goniometry, shape and texture identification (STI), Sollerman test, Disabilities of the arm, shoulder and hand questionnaire (DASH), two points discriminator and numeric pain scale
sensory threshold, range of motion, pain, function, tactile gnosia, pinch and grip strength | 6 months
  Semmes Weinstein monofilaments, Jamar® and Pinch Gauge® dynamometer, goniometry, shape and texture identification (STI), Sollerman test, Disabilities of the arm, shoulder and hand questionnaire (DASH), two points discriminator and numeric pain scale
sensory threshold, range of motion, pain, function, tactile gnosia, pinch and grip strength | 12 months
  Semmes Weinstein monofilaments, Jamar® and Pinch Gauge® dynamometer, goniometry, shape and texture identification (STI), Sollerman test, Disabilities of the arm, shoulder and hand questionnaire (DASH), two points discriminator and numeric pain scale

CONTACTS AND LOCATIONS:
Overall Officials: Marisa CR Fonseca, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Lucy Montoro Institute of Rehabilitation, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Result] Rosen B, Lundborg G. Training with a mirror in rehabilitation of the hand. Scand J Plast Reconstr Surg Hand Surg. 2005;39(2):104-8. doi: 10.1080/02844310510006187. PMID 16019738
- [Result] Rosen B, Lundborg G. Early use of artificial sensibility to improve sensory recovery after repair of the median and ulnar nerve. Scand J Plast Reconstr Surg Hand Surg. 2003;37(1):54-7. doi: 10.1080/alp.37.1.54.57. PMID 12625396
- [Result] Rosén B, Balkenius C, Lundborg G. Sensory re-education today and tomorrow: a review of evolving concepts. British Journal of Hand Therapy. v. 8, p. 48-56, 2003.
- [Result] Rosen B, Lundborg G. The long term recovery curve in adults after median or ulnar nerve repair: a reference interval. J Hand Surg Br. 2001 Jun;26(3):196-200. doi: 10.1054/jhsb.2001.0567. PMID 11386766
- [Result] Rosen B, Lundborg G. A model instrument for the documentation of outcome after nerve repair. J Hand Surg Am. 2000 May;25(3):535-43. doi: 10.1053/jhsu.2000.6458. PMID 10811759
- [Result] Rosen B, Lundborg G. A new tactile gnosis instrument in sensibility testing. J Hand Ther. 1998 Oct-Dec;11(4):251-7. doi: 10.1016/s0894-1130(98)80020-3. PMID 9862262
- [Result] Rosen B. Recovery of sensory and motor function after nerve repair. A rationale for evaluation. J Hand Ther. 1996 Oct-Dec;9(4):315-27. doi: 10.1016/s0894-1130(96)80037-8. PMID 8994006
- [Result] Rizzolatti G, Craighero L. The mirror-neuron system. Annu Rev Neurosci. 2004;27:169-92. doi: 10.1146/annurev.neuro.27.070203.144230. PMID 15217330
- [Result] Rizzolatti G, Fogassi L, Gallese V. Neurophysiological mechanisms underlying the understanding and imitation of action. Nat Rev Neurosci. 2001 Sep;2(9):661-70. doi: 10.1038/35090060. No abstract available. PMID 11533734
- [Result] Rizzolatti G, Luppino G. The cortical motor system. Neuron. 2001 Sep 27;31(6):889-901. doi: 10.1016/s0896-6273(01)00423-8. PMID 11580891
- [Result] Pons TP, Garraghty PE, Ommaya AK, Kaas JH, Taub E, Mishkin M. Massive cortical reorganization after sensory deafferentation in adult macaques. Science. 1991 Jun 28;252(5014):1857-60. doi: 10.1126/science.1843843.
- [Result] Orfale AG, Araujo PM, Ferraz MB, Natour J. Translation into Brazilian Portuguese, cultural adaptation and evaluation of the reliability of the Disabilities of the Arm, Shoulder and Hand Questionnaire. Braz J Med Biol Res. 2005 Feb;38(2):293-302. doi: 10.1590/s0100-879x2005000200018. Epub 2005 Feb 15. PMID 15785841
- [Result] Novak CB. Evaluation of hand sensibility: a review. J Hand Ther. 2001 Oct-Dec;14(4):266-72. doi: 10.1016/s0894-1130(01)80004-1. PMID 11762726
- [Result] Noble J, Munro CA, Prasad VS, Midha R. Analysis of upper and lower extremity peripheral nerve injuries in a population of patients with multiple injuries. J Trauma. 1998 Jul;45(1):116-22. doi: 10.1097/00005373-199807000-00025. PMID 9680023
- [Result] McAllister RM, Gilbert SE, Calder JS, Smith PJ. The epidemiology and management of upper limb peripheral nerve injuries in modern practice. J Hand Surg Br. 1996 Feb;21(1):4-13. doi: 10.1016/s0266-7681(96)80004-0. PMID 8676027
- [Result] Merzenich MM, Jenkins WM. Reorganization of cortical representations of the hand following alterations of skin inputs induced by nerve injury, skin island transfers, and experience. J Hand Ther. 1993 Apr-Jun;6(2):89-104. doi: 10.1016/s0894-1130(12)80290-0. PMID 8393727
- [Result] Ciechomska A, Kotwica Z. [Aphasia without alexia after surgical treatment of aneurysm of the right middle cerebral artery--incomplete lateralization of verbal functions?]. Neurol Neurochir Pol. 1991 Jul-Aug;25(4):516-20. Polish. PMID 1725057
- [Result] Lundborg G. Richard P. Bunge memorial lecture. Nerve injury and repair--a challenge to the plastic brain. J Peripher Nerv Syst. 2003 Dec;8(4):209-26. doi: 10.1111/j.1085-9489.2003.03027.x. PMID 14641646
- [Result] Lundborg G. Brain plasticity and hand surgery: an overview. J Hand Surg Br. 2000 Jun;25(3):242-52. doi: 10.1054/jhsb.1999.0339. PMID 10961548
- [Result] Lundborg G, Rosen B, Lindberg S. Hearing as substitution for sensation: a new principle for artificial sensibility. J Hand Surg Am. 1999 Mar;24(2):219-24. doi: 10.1053/jhsu.1999.0219. PMID 10194002
- [Result] Johansson BB. Brain plasticity in health and disease. Keio J Med. 2004 Dec;53(4):231-46. doi: 10.2302/kjm.53.231. PMID 15647628
- [Result] Jerosch-Herold C. Assessment of sensibility after nerve injury and repair: a systematic review of evidence for validity, reliability and responsiveness of tests. J Hand Surg Br. 2005 Jun;30(3):252-64. doi: 10.1016/j.jhsb.2004.12.006. PMID 15862365
- [Result] di Pellegrino G, Ladavas E, Farne A. Seeing where your hands are. Nature. 1997 Aug 21;388(6644):730. doi: 10.1038/41921. No abstract available. PMID 9285584
- [Result] di Pellegrino G, Wise SP. Visuospatial versus visuomotor activity in the premotor and prefrontal cortex of a primate. J Neurosci. 1993 Mar;13(3):1227-43. doi: 10.1523/JNEUROSCI.13-03-01227.1993. PMID 8441009
- [Result] di Pellegrino G, Fadiga L, Fogassi L, Gallese V, Rizzolatti G. Understanding motor events: a neurophysiological study. Exp Brain Res. 1992;91(1):176-80. doi: 10.1007/BF00230027. PMID 1301372
- [Result] Dellon AL, Jabaley ME. Reeducation of sensation in the hand following nerve suture. Clin Orthop Relat Res. 1982 Mar;(163):75-9. PMID 7067267
- [Result] Dagum AB. Peripheral nerve regeneration, repair, and grafting. J Hand Ther. 1998 Apr-Jun;11(2):111-7. doi: 10.1016/s0894-1130(98)80007-0. PMID 9602967
- [Result] Buccino G, Binkofski F, Riggio L. The mirror neuron system and action recognition. Brain Lang. 2004 May;89(2):370-6. doi: 10.1016/S0093-934X(03)00356-0. PMID 15068920
- [Result] Lundborg G. Nerve injury and repair - regeneration, reconstruction and cortical remodeling. Elsevier, Churchill Livingstone, 2a . ed. Cap.8, 9, 10 e 11, 198-244.
- [Result] LUNDBORG, G. Nerve injury and repair. Edinburgh, Churchill Livingstone, 1988.
- [Result] 9. HANSSON, T.; NYMAN, T.; NYLANDER, L.; ROSÉN, B.; BJÖRKMAN, A.; LUNDBORG, G. Visuell observation av taktil stimulering mot handen aktiverar sensomotoriska omraden I hjärnan. Svenska Läkaresällskapets Riksstämma. 2004. Abstract.
- [Result] DELLON, A.L.; Somatosensory testing and rehabilitation. The American Occupational Ther Ass, Inc. chapter:11, 246-293, 1997.
- [Result] DELLON, A.L. Evaluation of sensibility and re-education of sensation in the hand. Williams & Wilkins, 1981.
- [Derived] Paula MH, Barbosa RI, Marcolino AM, Elui VM, Rosen B, Fonseca MC. Early sensory re-education of the hand after peripheral nerve repair based on mirror therapy: a randomized controlled trial. Braz J Phys Ther. 2016 Jan-Feb;20(1):58-65. doi: 10.1590/bjpt-rbf.2014.0130. Epub 2016 Jan 19. PMID 26786080
- See also: School of Medicine - University of são Paulo — http://www.fmrp.usp.br